CLINICAL TRIAL: NCT04246723
Title: Efficacy and Safety of All-Oral Combination of Narlaprevir/Ritonavir and Sofosbuvir in Treatment-naïve Patients With Chronic Hepatitis C Genotype 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Almedis (Industry); Scientific Center EFiS (Unknown); ChromSystemsLab (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJ05013053
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Chronic Hepatitis c Genotype 1
Keywords: hepatitis; HCV; antiviral
MeSH Terms: conditions — Hepatitis | interventions — narlaprevir; Ritonavir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Narlaprevir + Ritonavir + Sofosbuvir for 12 weeks) (Experimental): All of enrolled patients receive equal study therapy with Narlaprevir 200 mg Once a day (QD)/Ritonavir 100 mg QD/Sofosbuvir 400 mg QD orally for 12 weeks. Narlaprevir should be taken with ritonavir and food and should be taken at approximately the same morning time each day.
  Sofosbuvir can be taken with or without meals.
  Interventions: Drug: Narlaprevir; Drug: Ritonavir; Drug: Sofosbuvir
- Cohort B (Narlaprevir + Ritonavir + Sofosbuvir for 8 weeks) (Experimental): All of enrolled patients receive equal study therapy with Narlaprevir 200 mg QD (once daily)/Ritonavir 100 mg QD/Sofosbuvir 400 mg QD orally for 8 weeks. Narlaprevir should be taken with ritonavir and food and should be taken at approximately the same morning time each day.
  Sofosbuvir can be taken with or without meals.
  Interventions: Drug: Narlaprevir; Drug: Ritonavir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Narlaprevir — 100 mg oval shaped, concave, yellow film-coated tablets taken as 200 mg per os once daily. 28 tabs/36 tabs/ 56 tabs in bottle.
Drug: Ritonavir — 100 mg tablets taken as 100 mg per os once daily. 30 tablets in bottle
Drug: Sofosbuvir — 400 mg yellow, capsule-shaped film-coated tablets debossed with "GSI" on one side and "7977" on the other side, taken as 400 mg per os once daily. 28 tablets in bottle.

SUMMARY:
Multicenter, open-label, phase II safety and efficacy study of all-oral combination of narlaprevir/ritonavir and sofosbuvir in Treatment-naïve Patients with Chronic Hepatitis C Genotype 1.

DETAILED DESCRIPTION:
Two patient cohorts were anticipated in this study:

1. Cohort A: 60 treatment-naive patients were enrolled into narlaprevir/ritonavir/sofosbuvir treatment for 12 weeks.
2. Cohort B: (exploratory): 25 treatment-naive patients with low viral load (HCV RNA<1000000 IU/L) were enrolled into narlaprevir/ritonavir/sofosbuvir treatment for 8 weeks.

The enrollment of 25 treatment-naïve patients with low viral load into 8 week cohort started after completion of enrollment of 60 treatment-naive patients into 12 week cohort.

The study included 3 time periods:

1. Screening period with duration up to 2 weeks during which study eligibility was confirmed.
2. Active treatment period (for 12 or 8 weeks): patients in the Cohort A were receiving study therapy with narlaprevir/ritonavir/sofosbuvir for 12 weeks, in the Cohort B - during 8 weeks.

   If a patient had virologic breakthrough while receiving therapy, discontinuation of antiviral treatment was advised with appropriate clinical follow-up.
3. Follow-up period during which patients did not receive any study medication. The duration of the follow-up period after the end of study treatment was 24 weeks.

Overall, each patient had been participating in the study for approximately up to 38 weeks from the time the patient signed the Informed Consent Form through the final visit.

If a patient had a screening failure, but was rescreened and subsequently enrolled, the reason for the original screening failure must have been documented in the source documents. A new subject Identification number (ID) was assigned to the patient.

The recruitment period in this study was planned to be up to 6 months. The total period of the study was anticipated to be approximately 1 year 3 months.

The patient was considered to be completed the study upon the completion of the last protocol specified visit. For those patients who did not complete the study, patient participation was considered terminated upon the completion of the last visit or contact (e.g., phone contact with the investigator).

It was estimated that 85 patients meeting inclusion/exclusion criteria would be recruited from approximately 6 clinical sites in Russia.

ELIGIBILITY:
Inclusion Criteria:

* Are willing and able to provide written informed consent.
* Have confirmed chronic HCV infection as documented by:

positive anti-HCV antibody (Ab) test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit

* Have HCV genotype 1 at screening as determined by the Central Laboratory. Any nondefinitive results must exclude the subject from study participation.
* Minimum HCV-RNA level of ≥ 10,000 IU at baseline;
* Treatment-naive patients to be enrolled into 8 week cohort must have HCV-RNA level <1,000,000 IU/L at baseline;
* No evidence of cirrhosis; availability at Baseline of at least one of the following tests negative results:

  1. Liver biopsy within 2 years of screening showing absence of cirrhosis
  2. Fibroscan® with a result of ≤ 12.5 kilopascal (kPa) within 6 months of baseline/Day1
  3. FibroTest® score of ≤ 0.48 AND Aspartate aminotransferase (AST)-to-Platelet Ratio Index (APRI) of ≤ 1 performed during screening

In the absence of a definitive diagnosis of the presence or absence of cirrhosis by the above criteria, a liver biopsy was required. Liver biopsy results supersede the results obtained by Fibroscan® or FibroTest®

* Have a screening electrocardiogram (ECG) without clinically significant abnormalities (P wave < 0.1 s; PQ interval 0,12-0,2 s; QRS complex 0,06-0,1 s; QT interval 0,35-0,49 s).
* Must have the following laboratory parameters at screening:

  1. alanine aminotransferase (ALT) ≤ 10 x the upper limit of normal (ULN)
  2. AST ≤ 10 x ULN
  3. Hemoglobin ≥ 12g/dL for male, ≥ 11g/dL for female subjects
  4. Platelets ≥ 50,000cells/mm^3 (for patients in 8-week study treatment group - ≥ 150,000 cells/mm3)
  5. International normalized ratio (INR) ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
  6. Albumin ≥ 3 g/dL;
  7. Direct bilirubin ≤ 1.5 x ULN;
  8. Hemoglobin A1c (HbA1c) ≤10%;
  9. Creatinine clearance (CLcr) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation.
* Have not been treated with any investigational drug or device within 30 days of the screening visit.
* A female subject is eligible to enter the study if it is confirmed that she is:

  1. Not pregnant or nursing;
  2. Of nonchildbearing potential (i.e., women who have had a hysterectomy, both ovaries removed, or medically documented ovarian failure, or are postmenopausal women >50 years of age with cessation [for ≥ 12 months ] of previously occurring menses), or
  3. Of childbearing potential (i.e., women who had not had a hysterectomy, both ovaries removed, or medically documented ovarian failure). Women ≤ 50 years of age with amenorrhea are considered to be of childbearing potential. These women must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the baseline/Day 1 visit prior to enrollment. They must also agree to one of the following from the screening until 6 months after last dose of the investigational drugs:

     * Complete abstinence from intercourse. Periodic abstinence from intercourse (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.
     * Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from the date of screening until 6 months after the last dose of the investigational drugs. Women of childbearing potential must not rely on hormone-containing contraceptives as a form of birth control during the study. Female subjects using a hormone-containing contraceptive prior to screening must stop their contraceptive regimen use from the date of screening until 6 months after their last dose of investigational drugs.
     * intrauterine device (IUD) with a failure rate of < 1 %;
     * female barrier method: cervical cap or diaphragm with spermicidal agent
     * tubal sterilization
     * vasectomy in male partner
* All male study participants must agree to consistently and correctly use a condom, while their female partner agrees to use either 1 of the nonhormonal methods of birth control listed above or a hormone-containing contraceptive listed below, from the date of screening until 6 months after their last dose of investigational drugs:

  * implants of levonorgestrel
  * injectable progesterone
  * oral contraceptives (either combined or progesterone only)
  * contraceptive vaginal ring
  * transdermal contraceptive patch
* Male subjects must agree to refrain from sperm donation for at least 6 months after the last dose of investigational drugs.
* Are in generally good health as determined by the investigator.
* Are able to comply with the dosing instructions for study drug administration and are able to complete the study schedule of assessments.

Exclusion Criteria:

* Had prior exposure to Interferon (IFN), ribavirin (RBV), or other approved or experimental Direct-acting Antivirals (DAA) targeting the HCV.
* Had prior exposure to amiodarone within 24 months before the screening
* Are pregnant or nursing female or male with pregnant female partner.
* Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, α1-antitrypsin deficiency, cholangitis).
* Are infected with hepatitis B virus (HBV) or human immunodeficiency virus(HIV).
* Have history of malignancy diagnosed or treated within 5 years; subjects under evaluation for malignancy are not eligible.
* Have chronic use of systemically administered immunosuppressive agents (e.g., prednisone equivalent > 10 mg/day).
* Have clinically relevant drug or alcohol abuse within 12 months of screening. A positive drug screen must exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by the investigator.
* Have excessive alcohol consumption, defined as more than 3 drinks on any single day and more than 7 drinks per week for females, and > than 4 drinks on any single day and more than 14 drinks per week for males.
* Have history of solid organ transplantation.
* Have history of clinically significant illness or any other major medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol by Investigators' opinion.
* Have history of a gastrointestinal disorder (or postoperative condition) that can interfere with the absorption of the study drug.
* Have history of difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
* Usage of any prohibited concomitant medications as described in the protocol (Appendix 1 - list of drugs with expected drug-drug interactions due to concomitant ritonavir usage)
* Have known hypersensitivity to the study investigational medicinal product, the metabolites, or formulation excipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieved Sustained Virologic Response (SVR12) in treatment-naïve patients cohort, received study therapy during 12 weeks. | Week 12 of follow-up period (SVR12) - week 24 of the study
  SVR12 - Undetectable HCV ( Hepatitis C Virus) RNA ( Ribonucleic Acid) by Lower limit Of Detection (LOD) 12 weeks following the end of treatment. LOD for HCV RNA <15 IU/mL

SECONDARY OUTCOMES:
The proportion of patients who achieved the Sustained Virological Response 24 weeks after the end of treatment (SVR24) in 12-week cohort | 24 weeks after the end of the treatment or week 36 of the study
  HCV RNA undetectable by LOD; for 12-week cohort patients
The proportion of patients achieved the End of treatment response (ETR) by LOD | Baseline and week 12 of the study (cohort A) or week 8 of the study (cohort B)
  HCV RNA <LOD at the treatment end;
The proportion of patients who achieved the Sustained Virological Response 4 weeks after the end of treatment (SVR4) by LOD | 4 weeks after the end of treatment - week 16 of the study for cohort A and week 12 of the study for cohort B
  HCV RNA <LOD 4 weeks after the end of treatment
The proportion of patients received 12 weeks of study treatment who developed viral breakthrough | week 12 of the study
  applicable for cohort A patients only; viral breakthrough defined as greater than or equal to 1 log10 increase in HCV-RNA above nadir, or detectable HCV-RNA, while on treatment after an initial drop below detection in 12-week cohort. Viral breakthrough is an unsatisfactory therapeutic effect. in this case discontinuation of antiviral treatment is advised with appropriate clinical follow-up. Viral breakthrough will be summarized by patient cohort and treatment regimen. The number and proportion of patients achieving undetectable HCV RNA at each time point will be summarized. Time to breakthrough will be estimated using the Kaplan - Meier method if applicable
The proportion of patients received 12 weeks of study treatment who developed relapse | week 12 of the study and week 24 of the study
  applicable for cohort A patients only; relapse presence is defined as HCV RNA undetectable by LOD at the end of treatment with subsequent detectable HCV RNA at the end of the follow-up period (week 12) in 12-week cohort;

OTHER OUTCOMES:
The proportion of treatment-naïve patients received 8 weeks of study treatment who achieve the SVR 12 by LOD | week 20 of the study
  HCV RNA <LOD
The proportion of patients received 8 weeks of study treatment who achieved SVR24 by LOD | week 32 of the study
  HCV RNA <LOD
The proportion of treatment-naïve patients received 8 weeks of study treatment achieved the ETR by LOD | Baseline and week 8 of the study (cohort B)
  HCV RNA <LOD at the treatment end;
The proportion of treatment-naїve patients received 8 weeks of study treatment who achieve the SVR4 by LOD | Baseline and week 12 of the study
  HCV RNA <LOD 4 weeks after the end of treatment;
The proportion of patients who develop viral breakthrough in treatment-naïve patients received 8 weeks of study treatment; | week 8 of the study
  applicable for cohort B patients only; viral breakthrough defined as greater than or equal to 1 log10 increase in HCV-RNA above nadir, or detectable HCV-RNA, while on treatment after an initial drop below detection in 12-week cohort. Viral breakthrough is an unsatisfactory therapeutic effect. in this case discontinuation of antiviral treatment is advised with appropriate clinical follow-up. Viral breakthrough will be summarized by patient cohort and treatment regimen. The number and proportion of patients achieving undetectable HCV RNA at each time point will be summarized. Time to breakthrough will be estimated using the Kaplan - Meier method if applicable
The proportion of patients who develop relapse in treatment-naïve patients received 8 weeks of study treatment. | week 8 of the study and week 20 of the study
  applicable for cohort B patients only; relapse presence is defined as HCV RNA undetectable by LOD at the end of treatment with subsequent detectable HCV RNA at the end of the follow-up period (week 12) in 8-week cohort;

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (5):
- Russia (5):
  - FBIS CSRI of Epidemiology of Federal Service on Customers, Moscow
  - FSIS FRC of food and biotechnology, Moscow
  - SBEI HPE MSMDU n.a. A.I. Evdokimov of Ministry of Health of Russia, Moscow
  - FSBI HEI HPE Military Medical Academy n.a. S.M. Kirov, Saint Petersburg
  - SPb SBIH Center on preventiomn and treatment of AIDS and infectional deseases, Saint Petersburg